CLINICAL TRIAL: NCT07027969
Title: Efficacy of Cardiometabolic Risk Factor Control Through Metabolic Surgery on Management and Severity of Atrial Fibrillation: METSAFE Randomized Clinical Trial
Brief Title: Metabolic Surgery for Atrial Fibrillation Elimination
Acronym: METSAFE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ali Aminian (Other)
Collaborators: Ethicon, Inc. (Industry); iRhythm Technologies, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ali Aminian, Director of Bariatric & Metabolic Institute, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-1039
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation; Obesity and Obesity-related Medical Conditions
Keywords: Atrial Fibrillation; Bariatric Surgery; Metabolic Syndrome; Weight Loss Surgery; Roux-en-Y gastric bypass; Sleeve Gastrectomy; GLP-1 Receptor Agonist; Tirzepatide; Semaglutide
MeSH Terms: conditions — Atrial Fibrillation; Obesity; Metabolic Syndrome | interventions — Gastric Bypass; Bariatric Surgery; Collagen Type II; Therapeutics

STUDY DESIGN:
Intervention Model Description: METSAFE is a randomized open-label blinded-endpoint single-center controlled efficacy/safety study with 2 parallel groups of patients with obesity and AF who will either receive metabolic surgery or nonsurgical obesity care for 30 months. The study has 2 phases: the first 12 months and the subsequent 18 months.
Masking Description: Patients and investigators will not be blinded to treatment assignment. However, the clinical assessors of cardiac rhythm recorders are blinded to the study arms; Assessment of the primary endpoint will be based on the blinded downloads and interpretation of Zio XT Patch (iRhythm) data yielding the AF burden.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metabolic Surgery (Active Comparator): Roux-en-Y Gastric Bypass (RYGB) and Sleeve Gastrectomy (SG)
  Interventions: Procedure: Roux-en-Y Gastric Bypass or Sleeve Gastrectomy
- Control group (nonsurgical standard of care for obesity) (Other): In the Control group, the subjects will be receiving standard of care for nonsurgical management of obesity, including possible AOMs that are not contraindicated in patients with AF at the discretion of obesity medicine specialists.
  Interventions: Drug: Anti-Obesity Medication (AOM) treatment

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass or Sleeve Gastrectomy — Patients receive either RYGB or SG. The surgical risk, differential impact of each procedure on body weight and other obesity-related diseases, presence of other medical and mental problems, patient's behavioral factors (e.g., postoperative compliance, active smoking), medications, and goals will be considered when the patient and local medical team make a shared decision about the most appropriate surgical procedure.
  Other Names: Roux-en-Y Gastric Bypass (RYGB); Sleeve Gastrectomy (SG); Bariatric Surgery
  Arms: Metabolic Surgery
Drug: Anti-Obesity Medication (AOM) treatment — Implementation of obesity pharmacotherapy in the nonsurgical group includes initial assessment of side effects and response, followed by achieving a clinically meaningful weight loss (5% weight loss) after three months. Once this goal is reached, AOMs will be continued throughout the study. If a weight plateau is reached within the first AOM, then another AOM may be added in combination in a stepwise fashion. The choice of AOMs considered may include metformin, topiramate, liraglutide, dulaglutide, semaglutide, tirzepatide, and empagliflozin.
  Arms: Control group (nonsurgical standard of care for obesity)

SUMMARY:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia. It is estimated that between 3 and 6 million Americans are currently living with AF, while 12 million people in the United States will have AF in 2030. Obesity and its comorbidities such as type 2 diabetes (T2DM), hypertension, and obstructive sleep apnea (OSA) are major risk factors for development and progression of AF. Metabolic and Bariatric Surgery (MBS) is the most effective currently available treatment for obesity. Patients typically lose 20 to 35 percent of body weight after surgery which is often sustained for many years. MBS can improve all 5 major risk factors of AF including obesity, hypertension, T2DM, OSA, and systemic inflammation.

The purpose of the study is to understand if MBS can affect the severity of AF and the toll AF's symptoms take on patients.

DETAILED DESCRIPTION:
This is randomized trial of 100 patients with BMI ≥35 kg/m2 and AF. Patients who met the initial screening criteria (including presence of at least 1% AF burden during a 2-week monitoring period with an ambulatory cardiac monitor) will be invited for possible enrollment. Patients will then be randomized 1:1 to MBS group versus nonsurgical control group and will be followed for 12 months (phase 1) and then for an additional 18 months (phase 2).

Interventions include Roux-en-Y Gastric Bypass or Sleeve Gastrectomy surgical procedures based on the shared medical decision between the bariatric surgeon and patients considering the patient's conditions. In the control group, patients are allowed to take anti-obesity medications (AOMs) that are not contraindicated in patients with AF at the discretion of obesity medicine specialists.

Lifestyle and risk factor modification in both groups will consist of targeted and personalized diet plans, exercise, and risk factor reduction, including optimal therapies for T2DM, hypertension, dyslipidemia, heart failure, coronary artery disease, and OSA.

ELIGIBILITY:
INCLUSION CRITERIA

Entry into the study would require that the patient:

1. Is a candidate for general anesthesia
2. Is eligible for metabolic surgery (RYGB or SG)
3. Is ≥18 and ≤80 years old
4. has a BMI ≥35 and ≤65 kg/m2
5. has AF criteria, which:

   1. Must be documented by EKG or cardiac monitor or Zio XT Patch
   2. Must have symptomatic AF
   3. In terms of types of AF, either paroxysmal AF with at least one episode lasting ≥5 minutes in the last 3 months prior to screening, or persistent AF, or longstanding AF.
   4. Must have a minimum burden of 1% during a 2-week screening time with an ambulatory noninvasive cardiac monitor.
   5. Must be assessed and confirmed by an expert cardiologist (e.g., cardiac electrophysiologist) to meet eligibility.
6. Patients without history of prior AF ablation/PVI procedure or with history of prior failed AF ablation/PVI procedure are eligible for the study.
7. Patients with and without T2DM are eligible for the study. Patients with T2DM should have been on a stable dose of anti-diabetic medication (including insulin) for at least 3 months prior to entry, with HbA1c ≤12%.
8. Have the ability and willingness to participate in the study and agree to any of the arms involved in the study.
9. Able to understand the options and to comply with the requirements of each arm.
10. Have a negative urine pregnancy test at screening and randomization visits for women of childbearing potential.
11. Women, of childbearing age, must agree to use reliable method of contraception for 2 years.

EXCLUSION CRITERIA

1. Significant cardiac valvular disease (planned to undergo cardiac valve intervention/surgery in the next 12 months)
2. Significant atherosclerotic disease (planned to undergo coronary, carotid, or peripheral artery revascularization procedures in the next 12 months)
3. Severe uncompensated cardiopulmonary disease leading to American Society of Anesthesiologists Class IV or V
4. Classified as New York Heart Association Class IV
5. Left ventricular ejection fraction <20% at the time of screening
6. Hospitalization for myocardial infarction, unstable angina, stroke, transient ischemic attack, heart surgery, coronary stent placement in the past 6 months
7. Prior bariatric and metabolic surgery of any kind (patients who had a gastric balloon or gastric band that were removed more than one year prior to enrollment are allowed to participate)
8. History of solid organ transplant
9. Type 1 diabetes or autoimmune diabetes
10. eGFR < 30 mL/min/1.73 m2 at screening or being on dialysis
11. Decompensated cirrhosis characterized by ascites, hepatic encephalopathy, portal hypertension, or esophageal varices.
12. Anemia defined as hemoglobin less than 9 g/dL
13. Use of investigational therapy
14. Liver transaminase level >300 U/L
15. Significant alcohol use (average >2 drinks/day)
16. Presence of active malignancy (except non-melanoma skin cancer)
17. Life expectancy less than 3 years due to concomitant diseases
18. Major mental health, psychological disorders, or substance abuse disorders that in the opinion of the investigators could disqualify the patient from metabolic surgery
19. Any condition or major illness that, in the investigator's judgment, places the subject at undue risk by participating in the study
20. Unable to understand the risks, benefits and compliance requirements of study
21. Lack capacity to give informed consent
22. Plans to move outside the primary location of study (Northeast Ohio) within the next 12 months
23. Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures
24. Known adhesive allergies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Relative change in total duration of being in atrial fibrillation (AF) | First 52 weeks of the study
  Relative change from baseline to 52 weeks in the percentage total duration of being in AF during a 2-week monitoring period (i.e., %burden), assessed by the Zio XT Patch (iRhythm).

SECONDARY OUTCOMES:
Presence of at least 1 AF episode | First 52 weeks of the study
  Presence of at least 1 AF episode (present or absent) in a 2-week monitoring time by Zio XT Patch at 52 weeks.
Change in number of AF episodes (≥30 seconds) | First 52 weeks of the study
  Change in Zio XT Patch derived variables from baseline to 52 weeks including number of AF episodes (≥30 seconds) in a 2-week monitoring time.
Change in number of AF espisodes longer than 6 minutes | First 52 weeks of the study
  Change in Zio XT Patch derived variables from baseline to 52 weeks including number of AF episodes longer than 6 minutes in a 2-week monitoring time.
Change in the longest AF duration | First 52 weeks of the study
  Change in Zio XT Patch derived variables from baseline to 52 weeks including the longest AF duration in a 2-week monitoring time.
Change in the second longest AF duration | First 52 weeks of the study
  Change in Zio XT Patch derived variables from baseline to 52 weeks including the second longest AF duration in a 2-week monitoring time.
Change in the AF type | First 52 weeks of the study
  Change in the AF type (e.g. regression from or progression to persistent form of AF)
Change in AF Symptom burden | First 52 weeks of the study
  Change in AF Symptom burden and severity assessed by the Toronto AF Severity Score (AFSS)
Relapse of AF after ablation | Throughout the study, 130 weeks
  Number of relapses of AF after ablation in each group
  *Since more ablation is expected in the second phase of study, this end point will be more relevant in the phase 2 of study.
Change in cardiac structure | First 52 weeks of the study
  Change in cardiac structure assessed by transthoracic echocardiography including LA and LV size, morphology, and function
Change in weight | First 52 weeks of the study
  Percent and absolute changes in body weight and BMI

OTHER OUTCOMES:
Percentage of Participants Achieving Weight Loss Milestones | First 52 weeks of the study
  Percentage of participants achieving ≥ 5%, ≥ 10%, ≥ 15%, ≥ 20%, ≥ 25%, ≥ 30%, ≥ 35% weight loss from baseline (yes/no)
Excess Weight Loss Percentage | First 52 weeks of the study
  Percentage of excess weight loss, calculated by dividing the difference between initial BMI and final BMI by the difference between initial BMI and a target BMI of 25
Change in waist circumference | First 52 weeks of the study
  Change in waist circumferential measurement above the level of the iliac crests measured in centimeters from baseline to 52 weeks
Change in physical activity | First 52 weeks of the study
  Change in physical activity, tracked by a commercial wearable device
Systolic blood pressure trends | First 52 weeks of the study
  Mean and change in systolic blood pressure in mmHg
Change in glucose homeostasis markers in T2DM patients | First 52 weeks of the study
  Mean and change from baseline in blood glucose and HbA1c in patients with T2DM
Percentage of patients with T2DM meeting predefined HbA1c targets | First 52 weeks of the study
  Percentage of patients meeting predefined HbA1c targets:
  * HbA1c <6.5% (without diabetes medications)
  * HbA1c <7% (irrespective of taking diabetes medications or not)
change in anti-diabetic medication | First 52 weeks of the study
  Changes in doses or drugs being used for diabetes
Mean and change from baseline in lipid panel | First 52 weeks of the study
  Mean and change from baseline in total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), and triglycerides
Changes in inflammatory markers (CRP) | First 52 weeks of the study
  Mean and change from baseline in C-Reactive Protein (CRP) in mg/L
change in antihypertensive therapy | First 52 weeks of the study
  Percentage of patients with escalation or de-escalation of antihypertensive therapy
change in antiarrhythmic therapy | First 52 weeks of the study
  Change in antiarrhythmic medications taken by the patient
Count of Direct Current cardioversions | First 52 weeks of the study
  Number of Direct Current (DC) Cardioversions
Count of AF ablation/pulmonary vein isolation procedures | Throughout the study, 130 weeks
  Number of AF ablation/pulmonary vein isolation (PVI) procedures (for increase in burden or persistence)
Other cardiovascular therapy changes | First 52 weeks of the study
  Change in other cardiovascular medications
Change in Quality of life metrics | First 52 weeks of the study
  Change from baseline in QoL metrics using Short Form Health Survey (SF-36)
Change in body composition (via Seca mBCA 554 Bioimpedance Analysis) | First 52 weeks of the study
  Change in body composition (% fat mass and % fat-free mass) as measured by Seca mBCA 554 Bioimpedance Analysis to examine correlation of changes in body composition with AF-related outcomes.
Change in Apnea-Hypopnea Index in polysomnoraphy | First 52 weeks of the study
  Change in Apnea-Hypopnea Index (AHI) in polysomnography to assess the possible positive effects of weight loss on OSA and to examine their correlation with AF-related outcomes
Count of major clinical outcomes | Throughout the study, 130 weeks
  Number of major clinical outcomes including all-cause mortality, cardiovascular mortality, stroke, transient ischemic attack, myocardial infarction, hospitalization for unstable angina, and hospitalization for heart failure.
Safety end points | Throughout the study, 130 weeks
  Complications specifically related to obesity, AF, metabolic surgery, as well as adverse events of cardiovascular medications and interventions in the trial will be recorded and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Aminani, Principal Investigator — Bariatric Research Medical Director
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No